CLINICAL TRIAL: NCT03649633
Title: Effect of Combined Vitamin C, Stress-dose Steroids, and Thiamine on Cerebral Autoregulation and Functional Outcomes of Patients with Septic Shock
Brief Title: Vitamin C, Steroids, and Thiamine, and Cerebral Autoregulation and Functional Outcome in Septic Shock
Acronym: CORVICTES-ΥΜ
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low rate of enrollment; publication of relevant results by other groups
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, Associate Professor of Intensive Care Medicine, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 163-10-5-2018
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Septic Shock
Keywords: Shock, Septic; Cerebrovascular Circulation; Spectroscopy, Near-Infrared; Patient Reported Outcome Measure
MeSH Terms: conditions — Shock, Septic | interventions — Ascorbic Acid; Placebo Effect

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, randomized, doubleblind, placebo-controlled, parallel-group clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroids/Vitamin C group (Experimental): "Combined Vitamin C and Stress-Dose Hydrocortisone": Patients with septic shock treated with 1500 mg Vitamin C every 6 hours for 4 days after randomization, and stress-dose hydrocortisone for 4 days (250 mg on day 1; and 200 mg on days 2, 3, and 4) after randomization.
  Interventions: Drug: Stress-dose Hydrocortisone plus Vitamin C
- Control group (Placebo Comparator): "Placebo plus placebo:" Patients with septic shock treated with placebo (corresponding to Vitamin C) and placebo (corresponding to hydrocortisone) for 4 days after randomization.
  Interventions: Drug: isotonic sodium chloride solution placebo plus isotonic sodium chloride solution placebo

INTERVENTIONS:
Drug: Stress-dose Hydrocortisone plus Vitamin C — Treatment of septic shock with vitamin C and stress-dose hydrocortisone aimed at the attenuation of the systemic inflammatory response and the improvement of vasopressor responsiveness.
  Other Names: Vitamin-Steroid
  Arms: Steroids/Vitamin C group
Drug: isotonic sodium chloride solution placebo plus isotonic sodium chloride solution placebo — Treatment of septic shock with placebo (corresponding to Vitamin C) and placebo (corresponding to hydrocortisone).
  Other Names: Placebo-placebo
  Arms: Control group

SUMMARY:
This study has been approved as a nested substudy of a multicenter trial (CORVICTES, Clinicaltrials.gov Identifier: NCT03592693). The current, randomized, placebo-controlled study will compare steroids/vitamin C versus placebo/placebo in septic shock, with respect to cerebral autoregulation, biomarkers, and functional outcome. The following hypotheses will be tested: The steroids/vitamin C/thiamine intervention may result in attenuation of the septic shock-associated impairment in cerebral autoregulation; and 2) The increased frequency of intact cerebral autoregulation in the intervention group may result in more neurologic failure free days and ventilator free days during a 60-day follow-up; improved survival to hospital discharge with good functional outcome; and better patient-reported health-related outcomes at 90-day follow-up.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Septic Encephalopathy is a serious complication of sepsis / septic shock. In postmortem, human brain samples, two forms of neuraxonal injury have been described, namely, scattered ischemic lesions and diffuse injury. Prior evidence suggests that cerebral autoregulation is impaired in patients with septic shock, and this may render the central nervous system more vulnerable to direct ischemic damage, especially during episodes of hypotension. Near-infrared spectroscopy (NIRS) constitutes an established method of noninvasive assessment of cerebral autoregulation and provides the capability of semiquantitative assessment of regional cerebral blood flow.

In the context of a multicenter randomized clinical trial (RCT) evaluating the effect of steroids and antioxidants on the outcome of septic shock, we aim to assess cerebral autoregulation and frontal cortex perfusion using NIRS in patients who will be enrolled in the 25-bed intensive care unit (ICU) of Evaggelismos Hospital, Athens, Greece.

The rationale of the main study is based on the following facts: A large body of experimental data has demonstrated that both corticosteroids and intravenous vitamin C reduce activation of nuclear factor kappa beta (NFƘB), thereby attenuating the release of pro-inflammatory mediators. This may result in reduced endothelial permeability and improved macrocirculatory flow, and augmentation of the release of endogenous catecholamines and enhanced vasopressor responsiveness. Furthermore, a combined attenuation of the systemic inflammatory response, reduced vascular leakage, and improved macrocirculatory flow may partly contribute to the preservation of cerebral autoregulation and effective, regional brain perfusion. In addition, recent evidence suggests that thiamine may be neuroprotective in severe shock states.

Regarding the rationale and hypotheses of the current substudy: Recent, observational data suggest that impaired cerebral autoregulation is independently associated with 3-month mortality in patients with septic shock. Therefore, the current project aims to test the following hypotheses: 1) The steroids/vitamin C/thiamine intervention may result in attenuation of the septic shock-associated impairment in cerebral autoregulation; and 2) The increased frequency of intact cerebral autoregulation in the intervention group may result in more neurologic failure free days and ventilator free days during a 60-day follow-up; improved survival to hospital discharge with good functional outcome; and better patient-reported health-related outcomes at 90-day follow-up.

METHODS

NIRS monitoring will be applied for 60 min at 2 levels of mean arterial pressure (MAP; ie, 65-70 mmHg and 95-100 mmHg) within 24-30 hours, and within 48-54 hours and 72-78 hours after the diagnosis of the septic shock. Autoregulation will be assessed by using tissue oxygenation index values and concurrently recorded MAP values in a regression analysis and will be considered as adequate if the pertinent Pearson correlation coefficient is lower than 0.3. Cerebral blood flow will be assessed by determination of the blood flow index after bolus injection of 5 mg of indocyanine green.

Patients will be randomized to the intervention or control group in subgroups of 4 using the "Research Randomizer" software, version 4 (https://www.randomizer.org/). Substudy intervention: In concordance with the main study protocol as approved by the Institutional Review Board (IRB; ie, the Scientific Council) of Evaggelismos Hospital, Athens Greece, the substudy intervention will comprise the following:

Hydrocortisone: Hydrocortisone 50 mg initial/single bolus (5-mL syringe containing 50 mg of hydrocortisone in normal saline), followed by a 24-hour continuous infusion of 200 mg/day for 4 days. The daily hydrocortisone dose of 200 mg will be diluted in a 50 or 100 mL bag of normal saline.

Hydrocortisone placebo will be provided as an identical syringe/50 or 100 mL bag of normal saline.

Vitamin C: Vitamin C is provided by the manufacturer as a 50 mL vial at a concentration of 500mg/mL. Three (3) ml of the vitamin C solution will be diluted in a 50 or 100 mL bag of normal saline (1500 mg vitamin C in a 50 mL bag) which will then be infused over 1 hour. The bag will be labeled by the study's pharmacy team as "vitamin C". The dosing schedule is 1500 mg every 6 hours for 4 days or until discharge from the ICU.

Vitamin C placebo will consist of an identical bag of 50 or 100 mL normal saline (but with no vitamin C) and will be labeled vitamin C. Placebo will be infused over 60 min as per the infusion instructions of the active vitamin.

Thiamine: As a high percentage of septic patients have been shown to be thiamine-deficient, patients will receive intravenous thiamine 200 mg every 12 hours for 4 days or until ICU discharge. Thiamine is also a cofactor for the metabolism of oxalate (a byproduct of vitamin C metabolism), with thiamine deficiency increasing oxalate levels. To simplify the study protocol both the intervention and the control group will receive thiamine.

The study inclusion and exclusion criteria are detailed in the dedicated subsections.

DOCUMENTATION AND PATIENT FOLLOW-UP

Monitoring of patients over the first 10 days after randomization will include: 1) Determination and recording of hemodynamic parameters and hemodynamic support, blood gases and fluid balance over the previous 24 hours as well as arterial blood lactate and central venous oxygen saturation; 2) Blood sampling at 24, 48 and 72 hours and 7 days after randomization for determination of cytokines' concentrations; 3) Daily, routine laboratory investigations' results and prescribed treatment data; 4) the results of 4 daily (1 / 6 hours) blood glucose measurements will be recorded and the incidence of hyperglycemia (defined as blood glucose over 200 mg/dL) will be analyzed; 5) Daily calculation of the Sequential Organ Dysfunction Assessment Score; and 6) The source of the infection, the results of blood cultures and other biological specimen cultures, and the antibiograms.

The time to first cessation of vasopressor support will also be documented. Follow-up until day 60 postresuscitation will include organ failure-free days and ventilator-free days. Finally, the ICU length of stay, the hospital discharge date, and the morbidity and complications / adverse events during hospital stay will be recorded.

ICU management protocol:

All septic patients enrolled in this study will be managed by a standardized approach which will comprise:

1. Empirical treatment with at least 2 broad spectrum antibiotics; antibiotic treatment will be deescalated according to microbiological data and clinical improvement
2. A conservative strategy of fluid management
3. A lung-protective ventilation strategy
4. Limited use of sedative agents according to pertinent guidelines
5. Enteral nutrition which will be started at 24 hours after ICU admission
6. Prophylaxis against deep venous thrombosis prophylaxis with both enoxaparin (or heparin in patients with a calculated creatinine clearance < 30 mL/min) and sequential compression/decompression stockings
7. Permissive hyperglycemia (ie, blood glucose of 150-200 mg/dL)

The study outcome measures are detailed in the dedicated subsection.

Sample size calculation: The previously reported frequency of impaired cerebral autoregulation is approximately 60% on day 2 after the diagnosis of sepsis/septic shock (3). The detection of a study intervention-related halving of the aforementioned proportion with an alpha value of 0.05 and a power of 0,80 would require the enrollment of 96 patients. As we estimate that at least 100 patients will be enrolled at Evagglismos hospital in the context of the steroids - vitamin C - thiamine multicenter RCT, we also propose a target enrollment of 100 patients for the current substudy.

G Power 3.1.9.2 Exact - Proportions: Inequality, two independent groups (Fisher's exact test) Options: Exact distribution Analysis: A priori: Compute required sample size Input: Tail(s) = Two Proportion p1 = 0.30 Proportion p2 = 0.60 α err prob = 0.05 Power (1-β err prob) = 0.80 Allocation ratio N2/N1 = 1 Output: Sample size group 1 = 48 Sample size group 2 = 48 Total sample size = 96 Actual power = 0.8004595 Actual α = 0.0290919

POSSIBLE SIGNIFICANCE OF STUDY RESULTS: In view of encouraging preliminary data on the corticosteroids / vitamin C, thiamine combination, we expect that the results of the current study will further elucidate important mechanisms underlying the (speculated) intervention-related benefit.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosis of septic shock within 12 hours of admission to the intensive care unit (ICU).

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Patients with a fatal underlying disease who are unlikely to survive to hospital discharge
* Patients with acquired immunodeficiency and a CD4 count of < 50 / μL
* Patients with known glucose-6 phosphate dehydrogenase (G-6PD) deficiency.
* Patients with sepsis/septic shock transferred from another hospital
* Patients with features of sepsis/septic shock > 12 hours
* Patients who require treatment with corticosteroids for an indication other than sepsis
* Patients with any history of an allergic reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Cerebral autoregulation | 24-78 hours after randomization
  Cerebral autoregulation while increasing MAP from a minimum of 65-75 mmHg to a maximum of 90-100 mmHg by changing the vasopressor infusion rate.
Cerebral blood flow | 24-78 hours after randomization
  Cerebral blood flow at an MAP of 65-75 mmHg and an MAP of 90-100 mmHg

SECONDARY OUTCOMES:
Neurologic failure free days | Days 1-60 after randomization
  Neurologic failure free days from day 1 to day 60 postrandomization; patients with a Glasgow Coma Scale Score of more than 9 will be considered as neurologic failure-free.
Ventilator-free days | Days 1-60 after randomization
  Ventilator-free days from day 1 to day 60 postrandomization; on any given follow-up day, patients will be considered as ventilator-free only in the absence of any need for ventilatory support within the preceding 24 hours.
Favorable, Inhospital, Neurological Outcome | Days 1-60 after randomization
  Survival to hospital discharge with a Cerebral Performance Category Score (CPC) of 1 or 2. The CPC score has 5 categories: 1 = good cerebral performance: the patient is conscious, alert, and able to work and lead a normal life; 2 = moderate cerebral disability: the patient is conscious and capable of independent activities of daily life; disorders such as hemiplegia, seizures, ataxia, cognitive changes, and/or noncerebral organ dysfunction causing moderate disability may be present; 3 = severe cerebral disability: patient is conscious and ambulatory but dependent on others, because of severe memory disturbance or dementia, or patient is paralyzed and can communicate only with his/her eyes, as in the locked-in syndrome; severe disability from noncerebral organ dysfunction may coexist; 4 = coma or vegetative state: patient is unconscious and unable of any verbal and/or psychological interaction with the environment; and 5 = death: certified brain death.
Patient-reported health-related quality of life: SF-36 | 90 days after randomization
  Patient-reported health-related quality of life by using the Short Form-36 Quality of Life questionnaire; available from: https://repository.niddk.nih.gov/static/studies/halt-pkd/Forms/F038%20Quality%20of%20Life.pdf; https://www.optum.com/campaign/ls/outcomes-survey-request.html.
  The Short Form 36 Quality of Life Questionnaire is a validated, 36-item, generic health status measure with scales of physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health, and reported health transition. The questionnaire is scored according to a norm-based scoring method. For example, assuming that an average normal person has a score of 50 in each scale, an individual respondent scoring below 45 is considered to have a "below-average" health status.
Biomarkers | 24-72 hours after randomization
  Plasma levels of tumor necrosis factor alpha (TNFa), interleukin (IL)-1 beta (1β), IL-6, IL-8, IL-10, Neuron Specific Enolase, and protein S100B at 24, 48, and 72 hours after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Spyros D Mentzelopoulos, MD, PhD, Principal Investigator — University of Athens Medical School; Anastasia Kotanidou, MD, PhD, Principal Investigator — University of Athens Medical School; Stylianos Orfanos, MD, PhD, Study Director — University of Athens Medical School; Spyros G Zakynthinos, MD. PhD, Study Chair — University of Athens Medical School
Locations (1):
- Evaggelismos General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
No specific plan